CLINICAL TRIAL: NCT06901466
Title: Strategies for Antithrombotic Treatment Following Transcatheter Edge-to-edge Repair in Patients With an Indication for Oral Anticoagulant: a Multicenter Randomized Controlled Trial
Brief Title: STrategies for AntithRombotic Treatment Following Transcatheter Edge-to-Edge Repair in Patients With an Indication for Oral Anticoagulant
Acronym: STAR-TEER Ⅰ
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-2612
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Mitral Regurgitation
Keywords: Transcatheter Edge-to-Edge Repair (TEER); Mitral Regurgitation; Cardiovascular Diseases; Embolism and Thrombosis; Bleeding; Aspirin; Rivaroxaban; Antithrombotic treatment; Oral anticoagulation; Platelet Aggregation Inhibitors; Stroke; Myocardial Infarction
MeSH Terms: conditions — Mitral Valve Insufficiency; Cardiovascular Diseases; Embolism and Thrombosis; Hemorrhage; Stroke; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban monotherapy (Experimental): Participants will receive rivaroxaban according to its indication within 12 months after the TEER. For patients using OAC at baseline, the OAC therapy is intended to be continued during perioperative period.
  Interventions: Drug: Experimental: Rivaroxaban monotherapy
- Rivaroxaban + Aspirin (Active Comparator): Participants will receive aspirin (100mg qd, 6 months) on top of rivaroxaban (according to its indication, 12months).For patients using OAC at baseline, the OAC therapy is intended to be continued during perioperative period.
  Interventions: Drug: Active Comparator: Rivaroxaban+Aspirin

INTERVENTIONS:
Drug: Experimental: Rivaroxaban monotherapy — Rivaroxaban monotherapy
  Arms: Rivaroxaban monotherapy
Drug: Active Comparator: Rivaroxaban+Aspirin — Rivaroxaban+Aspirin
  Arms: Rivaroxaban + Aspirin

SUMMARY:
Mitral regurgitation (MR) is the most common valvular heart disease, affecting approximately 24.2 million people worldwide (with a higher prevalence in older age groups). Transcatheter edge-to-edge repair (TEER) is now a well-established strategy in high-risk patients with MR. Globally, over 250,000 patients have benefited from the TEER technique.Studies have shown that patients with severe mitral regurgitation exhibit a high prevalence of atrial fibrillation (AF), reaching up to 63%, which is an indication for long-term oral anticoagulation (OAC) therapy. However, no dedicated study has prospectively evaluated different antithrombotic strategies following TEER in patients with an indication for OAC. Current guidelines do not provide any recommendations for the antithrombotic management of TEER. Consequently, considerable treatment variation exists in clinical studies and practice. The investigators will conduct a multicenter, open-label randomized trial to compare different antithrombotic strategies following TEER in patients who have an indication for OAC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone successful TEER (Defined as techinal success according to MVARC );
* Need for long-term oral anticoagulation;
* Ability to understand the requirements of the trial and willingness to comply with the trial protocol procedures;
* Providing written informed consent form；
* Women of childbearing potential must use an acceptable method of contraception from signing the informed consent form until the date of the last dose of antithrombotic drug;
* The heart team agrees on the antithrombotic strategies.

Exclusion Criteria:

* Severe renal impairment (creatinine clearance rate<15ml/min or on dialysis)；
* Postoperative persistent bleeding (overt bleeding either associated with a drop in the hemoglobin of 3.0 g/dl or requiring transfusion of 3 U of whole blood or packed red blood cells) or occurrence of vascular complications；
* Platelet count ≤ 30 ×10^9/L；
* Need for reoperation；
* History of intracranial or intracerebral hemorrhage；
* History of gastrointestinal ulcers or hemorrhage；
* Any hepatic disease associated with coagulopathy (Child-Pugh B or C);
* Allergy, intolerance or contraindication to oral anticoagulation or antiplatelet drug;
* History of cerebrovascular event or transient ischemic attack within the past 6 weeks;
* Current antiplatelet therapy；
* Patients who have participated in another drug or device investigational study within the past 30 days；
* Life expectancy <12 months；
* Pregnant or breastfeeding women。

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
All bleeding complications at 1 year after TEER | 1 year
  For the classification of bleeding complications, the Mitral Valve Academic Research Consortium (MVARC) Primary Bleeding Scale is used. All bleeding can be categorized into five types: minor bleeding, major bleeding, extensive bleeding, life-threatening bleeding, and fatal bleeding.

SECONDARY OUTCOMES:
Non-procedure-related bleeding complications at 1 year after TEER（key secondary outcome 1） | 1 year
  Non-procedure-related bleeding is consisted of all MVARC bleeding, excluding Bleeding Academic Research Consortium (BARC ) type 4 severe bleeding.BARC type 4 severe bleeding is defined by any of the following: perioperative intracranial bleeding within 48 hours, reoperation after closure of sternotomy for the purpose of controlling bleeding, transfusion of 5 or more units of whole blood or packed red cells within a 48-hour period, chest-tube output of 2 or more liters within a 24-hour period.
Composite of ischemic event (1)(key secondary outcome 2) | 1 year
  composite of all-cause mortality, stroke, systemic embolic events , or myocardial infarction at 1 year after TEER
Composite of ischemic event (2) | 1 year
  Composite of cardiovascular mortality, ischemic stroke, systemic embolic events ,or myocardial infarction at 1 year after TEER.
Composite of ischemic and bleeding events（1） | 1 year
  Composite of all bleeding, all-cause mortality, stroke, systemic embolic events or myocardial infarction at 1 year after TEER.
Composite of ischemic and bleeding events（2） | 1 year
  Composite of non-procedure-related bleeding events, cardiovascular mortality, ischemic stroke, systemic embolic events or myocardial infarction at 1 year after TEER.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Shouzheng Wang, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No